CLINICAL TRIAL: NCT05519098
Title: COLO-SW-1 Clinical Investigation
Brief Title: COLO-SW-1 Pivotal Clinical Investigation
Status: Completed | Type: Observational
Sponsor: Augere Medical AS (Industry)
Collaborators: Oslo University Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CIV-22-04-039386
Record Dates: First submitted 2022-08-23; First posted 2022-08-29 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Colonoscopy; Adenoma Colon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inclusion group: Patients referred for colonoscopy:
  * ≥18 years old
  * Consenting to participate
  Exclusion criteria:
  Endoscopists
  * Employment or family member employed at Augere Medical AS
  Patients:
  * Severe comorbidity, NYHA III-IV
  * Pregnancy
  * Hospitalized patients
  * Active inflammatory bowel disease
  * Poor bowel preparation defined as Boston Bowel Preparation Score as ≤1 in any segment
  * Absence or unable to provide consent
  * Cecum not reached
  Interventions: Device: COLO-SW-1

INTERVENTIONS:
Device: COLO-SW-1 — Patient will undergo a CADe-assisted colonoscopy procedure with use of the COLO-SW-1 software.

SUMMARY:
The Clinical Investigation is a summative usability study and a 'first-in-patient'-study of the independent medical device software (MDSW) utilizing artificial intelligence. The MDSW has completed the development phase and is ready to enter production. The primary objective of this study is to assess the user safety and secondary the user-friendliness of the MDSW to confirm compliance to certain General safety and performance requirements (GSPR) set by the MDR. The software to assess will be installed in a medical grade PC to allow the use of the MDSW according to its intended purpose of detecting colorectal polyps. However, the PC is not a part of the medical device under investigation and its performance and safety will not be assessed by this investigation. The intended purpose and clinical benefit of the MDSW is to assist the endoscopist in detecting more polyps, with the possibility of subsequently preventing colorectal cancer later on. The data obtained from the investigation will be used for regulatory purposes aiming to obtain a CE certification as class IIa according to MDR for the MDSW under investigation.

The multi-center investigation will assess 8-20 endoscopists experience with the MDSW and whether technical difficulties occur during its use in one site. The user experience of the endoscopists will be collected in a questionnaire form. The investigator will additionally record any possible adverse effects (AE) or adverse technical effects (ATE) of the use of the MDSW. The MDSW will be used during ordinary colonoscopy in adult, out-patients ≥18 years but variables related to the patient outcome will not be assessed. Patients with inadequate bowel preparation, active inflammation, cecum not reached or not consenting will be excluded from the study. Each endoscopist will assess the device during 3-5 patient examinations.

The primary objective of the investigation is to confirm that COLO-SW-1 is safe for use during colonoscopy as intended for aiding in detection of polyps. The secondary objective is to assess the user-friendliness of the MDSW interface.

The clinical investigation is estimated to start in August 2022. The participation of the endoscopists will take place continuously through the clinical investigation until required number (up to 20) of participants has been reached. When 8 participants have been included in total, an interim analysis is made, and the Principal Investigator decides if the confirmatory objectives have been met. A conclusion can be drawn from the partial objectives met at this point. The study can continue for up to 20 participants to complete all endpoints, if required. The investigation will be closed by end of October 2022. The investigation will be deemed completed once the last evaluation form has been completed by the endoscopists.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Consenting to participate

Exclusion Criteria:

* Severe comorbidity, NYHA III-IV
* Pregnancy
* Hospitalized patients
* Active inflammatory bowel disease
* Poor bowel preparation defined as Boston Bowel Preparation Score as ≤1 in any segment
* Absence or unable to provide consent
* Cecum not reached

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population with a referral to colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AE) | 2 months
Number of technical problems disturbing the colonoscopy | 2 months
  1. Artifacts in the images on the endoscopy monitor
  2. Degradation of the endoscopic image quality due to the device
Confirming compatibility to the endoscopic system | 2 months
  The outcome is assessed by user questionnaire

SECONDARY OUTCOMES:
User manual understandability | 2 months
  The outcome is assessed by user questionnaire
Ease of activation of the device | 2 months
  The outcome is assessed by user questionnaire
Quality of visual alert | 2 months
  The outcome is assessed by user questionnaire
If the visual overlay disturbed polyp characterization | 2 months
  The outcome is assessed by user questionnaire
Number of procedures used with an AI system, the one under the investigation | 2 months
  The outcome is assessed by user questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Oslo University Hospital, Oslo, Norway
- Sahlgrenska University Hospital-Mölndal, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No